CLINICAL TRIAL: NCT04478812
Title: A Prospective, Multi-Center, Blood Collection Study to Evaluate TbitTM System Precision and Correlation Between Different Blood Samples Measured With TbitTM System
Brief Title: Tbit System Precision and Correlation of Different Blood Samples
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioDirection Inc (Industry)
Responsible Party: Sponsor
Organization: NanoDx (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BDI-TBIT-04
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Brain Injuries; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Group Assignment (Experimental)
  Interventions: Diagnostic Test: Single Group Assignment

INTERVENTIONS:
Diagnostic Test: Single Group Assignment — Tbit™ System will detect S100B and GFAP concentrations with the blood specimen collected

SUMMARY:
The Tbit™ System will detect S100B and GFAP concentrations with the blood specimen to produce and compare repeated measures from 3 blood samples from 3 fingersticks from one subject and one 1 venous whole blood sample will be collected from the same subject, on 3 different Tbit™ System by 3 different operators.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Presents to the Emergency Department with suspected traumatic brain injury
* Blood sample collected for Tbit™ System within 12 hours of injury
* Willing and able to provide informed consent or obtain consent from legal authorized representative (LAR)

Exclusion Criteria:

* Suspect of ischemic or hemorrhagic stroke with subsequent incidental trauma based on ED examination
* Subject suspect of need of craniotomy for the acute trauma for this event
* External signs compatible with a depressed skull fracture based on ED exam
* Subject requiring administration of blood transfusion after injury and prior to study blood draw
* Subject for whom timing of injury is unable to be estimated within 1 hour of certainty
* Subject who had neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizures, brain tumors, stroke or TIA within the last 30 days, or history of neurosurgery
* Known or suspected to be pregnant
* Prisoner or under incarceration
* Participating in another clinical research study prior to this study completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Measurement Repeatability | within 12 hours from injury for Tbit and within 30 min from the sample drawn
  1. Evaluate the repeatability of measurement of S100B and GFAP concentrations in capillary blood using the Tbit™ System at different clinical sites and between-instrument and between-operator components of variance in the intended use environment.
Compare Measurements | within 12 hours from injury
  2. Compare concentrations of S100B and GFAP measured using Tbit™ System in specimens obtained from a fingerstick blood, venous whole blood, serum and plasma in the intended use environment.

CONTACTS AND LOCATIONS:
Overall Officials: Jerika Acosta, BSc, Study Director — Medicept Inc.

IPD SHARING:
Plan to Share IPD: Undecided